CLINICAL TRIAL: NCT06352333
Title: Parasagittal Vs Cornerpocket Approaches for Ultrasound Guided Supraclavicular Brachial Plexus Block A Comparative Study
Brief Title: Parasagittal Vs Cornerpocket Approaches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nada Thabet Ahmed, Principle investigaror, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Parasagittal Vs Cornerpocket
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Supraclavicular Brachial Plexus Block
Keywords: brachial plexus block

STUDY DESIGN:
Intervention Model Description: Inclusion criteria:
  * 18to60 yearsold
  * ASA grade I to II
  * Elective upper limb surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Cornerpocket supraclavicular ultrasound guided brachial plexus block
  Interventions: Procedure: supraclavicular ultrasound guided brachial plexus block
- group B (Active Comparator): Parasagital supraclavicular ultrasound guided brachial plexus block
  Interventions: Procedure: supraclavicular ultrasound guided brachial plexus block

INTERVENTIONS:
Procedure: supraclavicular ultrasound guided brachial plexus block — two approaches of ultrasound guided supraclavicular brachial plexus block in upper limb surgery : the cornerpocket supraclavicular brachial plexus block and parasagittal supraclavicular brachial plexus block

SUMMARY:
Brachial plexus blocks are widely used to provide anesthesia for upper limb surgery.

Although many different approaches to the brachial plexus block have been described, there is widespread acceptance that injecting at the supraclavicular level is the most reliable method in terms of spread of local anesthetic agent.

Each approach of ultrasound guided supraclavicular brachial plexus block (US -SCBPB ) has a different success rate and complications. .

A supraclavicular block can provide effective surgical anesthesia of the forearm and hand.

The most commonly performed US- SCBPB is the corner pocket approach which was described by Chan et al with probe resting posterior to the clavicle, with postero latero-anteromedial orientation provides a very stable location, but has the disadvantage of "looking" across the first rib, with the apex of the lung visualized close to thePlexus .

A new Parasagittal approach for brachial plexus block at the supraclavicular level was studied by Adrian Searle where the arc of the first rib was used to provide a deep limit to needle transit in order to minimize the risk of pneumothorax ;the aim of our study is to further evaluate the parasagittal approach for brachial plexus block and compare it with the popular corner pocket approach

DETAILED DESCRIPTION:
After approval of research ethics committee of Sohag University hospital, a written consent will be taken from all participants to use their data for research and educational purposes The study will be carried on 80 participants who undergo elective upper limb surgery for a comparative study.

In this study the investigators will use A 22 G Spinal needle , a high frequency linear probe of US and 2 % lidocaine and 0.5% bupivacaine as local anathetics ,Every participant will be informed about advantages and disadvantages of the research and has the right to withdraw at any stage without negative impact on medical service production.

For both types of block:

Wide bored cannula is inserted,Monitoring is applied (pulse,Ecg,Bp) Oxygen mask 5 liters , Participants were positioned supine with the head turned to the non-operative Side ( contralateral side), and a pillow under the head and shoulder with the ipsilateral arm placed adducted by the patient side.

After that we sterilize the skin and apply a local anesthetic (2-3 ml of2% lidocaine).

The total volume of the local anesthetic mixture was 30 ml (10 ml of 2% lidocaine mixed with 20 ml of 0.5% bupivacine ) Then participants will be divided randomly into 2 groups ,each group 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old
* ASA grade I to II
* Elective upper limb surgery

Exclusion Criteria:

* Patient refusal.
* Patient with neurological deficit in the limb of surgery
* Patients with psychiatric disease.
* Coagulopathy.
* Morbid obesity.
* Known allergy to used local anathetics
* Local infection at the block site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Needle visibility in both approaches | 1 year
  Measure the visibility of the needles in the ultrasound

SECONDARY OUTCOMES:
Duration of sensory and motor block | 1 year
  Measure the time of sensory and motor block start to happen after injecting local anathetics

OTHER OUTCOMES:
Success rate | 1 year
  Measrue number of failed and successful nerve blocks
Complications | 1 year
  Measure complications of the block

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Choi S, McCartney CJ. Evidence Base for the Use of Ultrasound for Upper Extremity Blocks: 2014 Update. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):242-50. doi: 10.1097/AAP.0000000000000155. PMID 25376973
- [Background] Soares LG, Brull R, Lai J, Chan VW. Eight ball, corner pocket: the optimal needle position for ultrasound-guided supraclavicular block. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):94-5. doi: 10.1016/j.rapm.2006.10.007. No abstract available. PMID 17196502
- [Background] Chan VWS, Perlas A, Rawson R, Odukoya O. Ultrasound-guided supraclavicular brachial plexus block. Anesth Analg. 2003 Nov;97(5):1514-1517. doi: 10.1213/01.ANE.0000062519.61520.14. PMID 14570677
- [Background] Duggan E, El Beheiry H, Perlas A, Lupu M, Nuica A, Chan VW, Brull R. Minimum effective volume of local anesthetic for ultrasound-guided supraclavicular brachial plexus block. Reg Anesth Pain Med. 2009 May-Jun;34(3):215-8. doi: 10.1097/AAP.0b013e31819a9542. PMID 19587618